CLINICAL TRIAL: NCT06136468
Title: Understanding the Impact of Humanoid Technology (HT) Driven Health Enhancing Physical Activity (HEPA) Program Among Community-Dwelling Filipino Older Adults
Brief Title: Humanoid-Technology Driven Health Enhancing Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00347131
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Community-dwelling Older Adults
Keywords: Health enhancing physical activity; Virtual coach

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Exercise program using the "virtual coach" projected through head-mounted display
  Interventions: Behavioral: Virtual coach
- No Intervention (No Intervention): Usual exercise program

INTERVENTIONS:
Behavioral: Virtual coach — The virtual coch will be displayed to the participants using an optical see-through head-mounted display
  Arms: Experimental

SUMMARY:
Ensuring the health and well-being of older individuals is a global problem. The application of emerging technology is increasingly advocated to improve health outcomes, yet the investigators need to identify how feasible and acceptable this is among users. One example of these emerging technologies is humanoid technologies. Humanoid technologies are human-resembling digital objects that can be projected using head-mounted displays to be worn by users. This study seeks to assess the impact of humanoid technologies (HTs) in the form of digital health coaches to enhance the physical activity of community-dwelling older adults in the Philippines. The quasi-experimental study will assess the participants' intention for technology use and the participants experience of the intervention (acceptability, barriers, and facilitators). Specifically, this study will compare the impact of the Humanoid Technology-driven Health Enhancing Physical Activity program versus a standard physical activity program (video-based) on physical performance, cognitive function, and quality of life among older adults in two 'senior centers' in the Philippines. The study will also identify older adults' preferences for an ideal Humanoid Technology-driven Health Enhancing Physical Activity and the participants intention to use it via survey. An embedded qualitative study will explore participants' perceptions of the acceptability, barriers, and facilitators of the Humanoid Technology-driven Health Enhancing Physical Activity program.

DETAILED DESCRIPTION:
A quasi-experimental research design with embedded qualitative interviews will be used to understand the impact of Humanoid Technology-driven Health Enhancing Physical Activity among community-dwelling Filipino older adults and compare the effects of Humanoid Technology-driven Health Enhancing Physical Activity versus the current Health Enhancing Physical Activity (live coaching and video-based) on the participants' physical, cognitive status, and Quality of Life.

The investigators will assess the preferences of the older adults prior to the intervention to identify the participants specific wishes and choices (e.g., music, gender of the humanoid technology coach). To achieve this, the investigators will follow the conjoint analysis methods in healthcare as follows: (a) defining intervention attributes and levels based on literature evidence and (b) designing the attributes and levels as components of the program, and (c) designing the conjoint survey questionnaire. The computer-based survey questionnaire using the Sawtooth software will be distributed to participants.

The investigators have identified two community senior centers affiliated with the local government unit to participate in this quasi-experimental study. One community senior center will serve as the experimental site and the second community senior center will serve as the control site. Older adults will be recruited at each site for study participation.

The eligible participants will be purposively selected from the regular attendees at the study sites using the inclusion criteria: (1) ambulatory, (2) can follow simple instructions, (3) normal eyes functioning without low vision (or at most with corrective lenses), and (4) willingness to participate in the program with signed informed consent. Older adults who are considered not suitable to participate by the community physician using the local guidelines will be excluded. A total of 128 or 64 older adults in each center, will be recruited via posters at community senior centers. Afterward, the treatments will be assigned to each of the two senior center sites for the quasi-experimental study. Only the participants from the experimental group shall be involved in the usability evaluations and six from the experimental group for the qualitative study.

The intervention period will run for 1 month consisting of the first two weeks of the twice-weekly (Tuesday and Thursday) schedule to be followed by the second 2 weeks of three times weekly (Monday, Wednesday, Friday) schedule. Each session will last approximately 1.5 hours, including orientation, warm-up, and stretching. All participants will be supervised by the health team and trained personnel at the senior center and follow a standard protocol. The investigators will compare the participants physical, cognitive status, and Quality of Life measures before and after the intervention using standardized methods.

After the intervention, the investigators will ask the older adults in the experimental group to answer a survey related to the usability of the program and the participants intention to participate in the program in the future. The investigators will select six participants from the experimental group for an interview to know the participants perception of the intervention, particularly related to its acceptability, barriers, and facilitator.

As with other studies involving technologies, potential risks include loss of autonomy, privacy, data protection, safety, isolation prevention, and user over-stressing. To minimize the risks, proper orientation will be held. The research team will undergo training and acquire good clinical practice certificate. Procedures will align with the currently accepted standards by the (local) Philippine Department of Health, the research team will recruit social workers and healthcare providers to monitor the interventions and for potential health and wellness issues during the study. Reporting untoward events will comply with the current protocol and standards.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory
* can follow simple instructions
* normal eyes functioning without low vision (or at most with corrective lenses), (4) willingness to participate in the program with signed informed consent

Exclusion Criteria:

* non-ambulatory
* not suitable to participate as certified by a community physician

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-10-14 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Change in Physical Status as assessed by the 6 minute walk test | baseline; 2 weeks, 4 weeks
  6-minute walk test
Change in Cognitive Status as assessed by the Montreal Cognitive Assessment (MoCA) | baseline; 2 weeks, 4 weeks
  Montreal Cognitive Assessment, 0-30 scores, higher scores mean a better outcome
System Usability as assessed by the Post Study System Usability Questionnaire | after intervention up to 1 week
  Post Study System Usability Questionnaire measure is scored on a 0-100 scale, and a higher score means a better outcome. This questionnaire contains 16 items on a 7-point likert.
Technology Acceptance as assessed by the Unified Theory of Acceptance and Use Technology (UTAUT) Questionnaire | after intervention up to 1 week
  Unified Theory of Acceptance and Use Technology (UTAUT) Questionnaire is a 8-construct, 31-item questionnaire. The items are measure along a 7-point Likert scale, which ranges from "strongly agree" (1) to "strongly disagree" (7)
Change in Health related quality of life as assessed by the Short Form 8 (SF-8) Questionnaire | baseline; 2 weeks, 4 weeks
  SF-8 Questionnaire is a 2-construct, 8-item questionnaire assessing mental and physical health scores which is measures using 6 point scale: (0) Poor to (6) Excellent

SECONDARY OUTCOMES:
Health behavior | baseline
  Health behavior as assessed by Patient Action Inventory for Self-Care. It consists of 57 items. Participants were asked to indicate Yes or No for each action statement from three perspectives: 1) Is this important to you? 2) Do you want to do this? 3) Are you able to do this?. For each action item, the mean value will be used to describe the percentage of the participants answered Yes as 1 versus No as 0; and 2) by each of the three perspectives - importance, desirability, and perceived ability. The ranks are indicated from the highest to the lowest percentage, where Rank 1 indicates the item that most participants indicated with Yes. The arithmetic mean will be used as a measure of importance, desire, and ability levels for each action item.
Geriatric Depression as assessed by Geriatric Depression Scale | baseline
  The Geriatric Depression Scale (GDS) is a 15-item self-report measure of depression in older adults where subjects respond in a Yes/No format. Out of the 15 items, 10 indicate the presence of depression when answered positively, while the other 5 are indicative of depression when answered negatively. The form can be completed in approximately 5 to 7 minutes, making it ideal for people who are easily fatigued or are limited in their ability to concentrate for more extended periods of time.
Sleep Quality as assessed by Pittsburgh Sleep Quality Index | baseline
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances. The score ranges from 0-21. Scores higher than 5 indicate poor sleep quality.
Anxiety Symptoms as assessed by Spielberger State-Trait Inventory (STAI) | baseline
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Demographics and Literacy as assessed by researcher-made questionnaire. | baseline
  Consists of residence, gender, age, marital status, education, and self-rated technology literacy/competency and general health

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Himmelfarb, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- Philippines (2):
  - Quezon City Senior Citizens Affairs, Quezon City, NCR
  - Valenzuela Senior Citizens Affairs, Valenzuela, NCR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dino MJS, Dion KW, Abadir PM, Budhathoki C, Balbin PT, Malacas MKG, Hernandez RP, Nicolas JJG, Barcial-Espinosa J, Himmelfarb CRD, Davidson PM, Thiamwong L. Community-Dwelling Filipino Older Adults' Experiences with Virtual Coach for Health-Enhancing Physical Activity (HEPA): A Phenomenology. Nurs Rep. 2025 Jan 31;15(2):49. doi: 10.3390/nursrep15020049. PMID 39997785
- [Derived] Dino MJS, Dion KW, Abadir PM, Budhathoki C, Huang CM, Padula WV, Himmelfarb CRD, Davidson PM. The impact of a mixed reality technology-driven health enhancing physical activity program among community-dwelling older adults: a study protocol. Front Public Health. 2024 May 14;12:1383407. doi: 10.3389/fpubh.2024.1383407. eCollection 2024. PMID 38807990